CLINICAL TRIAL: NCT01699867
Title: Computed Optical Margin Assessment for Breast Cancer Surgery, Phase I (Part A)
Status: Completed | Type: Observational
Sponsor: Diagnostic Photonics, Inc. (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: DxP 2012-02 (Part A)
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: lumpectomy; breast cancer; optical coherence tomography; tumor margin; imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Optical coherence tomography — Optical coherence tomography was used to image ex vivo breast tissue specimens.

SUMMARY:
This multi-center, prospective, open label study analyzed specimens from fifty subjects at two study sites. Patients scheduled to undergo breast-conserving surgery were recruited in accordance with the inclusion and exclusion criteria. The study period per subject was the time it took to assess the ex vivo breast tissue sample using the study device. Image review was conducted after surgery and compared to the margin status findings in the post-operative pathology report.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years of age or older
2. Signed informed consent form
3. Women who have been histologically diagnosed with carcinoma of the breast prior to surgery
4. Patients planning breast preservation and undergoing lumpectomy (partial mastectomy) procedure

Exclusion Criteria:

1. Multicentric disease (histologically diagnosed cancer in two different quadrants of the breast)
2. Neoadjuvant systemic therapy
3. All T4 tumors
4. Previous radiation in the operated breast
5. Prior surgical procedure in the same quadrant
6. Implants in the operated breast
7. Pregnancy
8. Lactation
9. Participating in any other investigational study for either drug or device which can influence collection of valid data under this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer undergoing lumpectomy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa K Jacobs, M.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Optical Coherence Tomography (Single-arm): Specimens from all patients were evaluated by optical coherence tomography.
Period: Overall Study
Arm/Group | Optical Coherence Tomography (Single-arm)
Started | 50
Completed | 47
Not Completed | 3
Not completed — Screening Failure | 3

BASELINE CHARACTERISTICS:
Population: 47 patients completed the study. 1 patient was excluded from the analysis due to insufficient images in all specimens (did not meet protocol specifications).
Arm/Group | Optical Coherence Tomography (Single-arm)
Number analyzed (Participants) | 46
Age, Continuous [Mean (Full Range); unit: years] | 62 [27 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Patients With All Positive Margins Correctly Identified With the Device
Description: In this study, a patient had "positive margins" if tumor was identified at the true margin (i.e., the final margin or new margin) surface of at least one specimen by histology (0 mm, "tumor on ink").
Time Frame: one week after surgery
Population: Patients with positive margins (0 mm, "tumor on ink").
Measure: Number; unit: Patients w/ all positives identified
Arm/Group | Optical Coherence Tomography (Single-arm)
Number analyzed (Participants) | 8
Patients w/ all positives identified | 5

2. Primary Outcome: Number of Margins With False Positive Device Readings
Time Frame: one week after surgery
Population: Patients with all negative margins (≥ 2 mm). On average, 5 out of 6 possible margins were analyzed per patient.
Measure: Mean (Standard Deviation); unit: False positive margins per patient
Arm/Group | Optical Coherence Tomography (Single-arm)
Number analyzed (Participants) | 35
False positive margins per patient | 1.32 (1.38)

ADVERSE EVENTS:
Time Frame: During the surgical procedure.
Description: The investigational device only contacted excised patient tissue. The device did not contact patients as part of this study.
Groups:
- All Patients (Single-arm): All enrolled study patients.
Arm/Group | All Patients (Single-arm)
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No